CLINICAL TRIAL: NCT06726408
Title: Critical Care Optimized Pediatric Quantitative EEG
Brief Title: Critical Care Optimized Pediatric and Neonatal Quantitative Neuromonitoring
Acronym: COPeQ
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0381; N° ID-RCB : 2024-A01607-40 (Other: Agence nationale de sécurité du médicament et des produits de santé (ANSM))
Record Dates: First submitted 2024-11-28; First posted 2024-12-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Intensive Care Unit
Keywords: Quantitative neuromonitoring; Pediatric and neonatal critical care; Neonatal encephalopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neuromonitoring with 10 electrodes — In case of no parental objection, the clinician may begin neuromonitoring according to standard indications. The number of electrodes applied to the child's skull will be 10 electrodes (8 recording electrodes, 1 reference electrode, and 1 ground electrode) instead of the current 5.
  The intensivist will analyze the quantitative EEG trace as they currently do but will also have access to additional tools for seizure detection support (CDSA and seizure detection software) and targeted review of part of the recording by a neurophysiologist in case of doubt. Access to the neurophysiologist will be available during current working hours on weekdays. Data will be collected in 12-hour periods.

SUMMARY:
The detection and appropriate treatment of seizures significantly impact the neurological prognosis of patients in intensive care. Indeed, altered brain function including seizures is described in critically ill children, regardless of the reason for admission. Most seizures are subclinical and therefore impossible to diagnose without neuromonitoring tools. Despite being concidered ad Gold Standard, continuous EEG (cEEG) with video recording shows difficulty of implementation and interpretation at all hours of the day and night explaining that less than 10% of centers in France use cEEG routinely. Most departments prefer simplified techniques, including amplitude traces (aEEG) which can be used continuously at the bedside. However, the positive predictive value of aEEG in the detection of seizures does not exceed 78% and 64% in newborns and children respectively making necessary an optimization of the information provided by these techniques.

This project is a pragmatic diagnostic study that aims at developing and evaluating a neuromonitoring interface adapted to the needs of pediatric and neonatal intensive care units and meeting the requirements of neurophysiologists in terms of EEG trace quality.

DETAILED DESCRIPTION:
This research will take place in three phases :

1. Parameterization of the interface, which will display an 8-channel aEEG trace associated with reading aids (CDSA and automated seizure detection) available to the clinician.
2. Teams' training regarding the placement of additional electrodes and the use of reading aid tools.
3. Patient's inclusion. The obtained traces will be accessible at any time for direct interpretation and can be read on demand by a neurophysiologist during office hours.

Post-hoc review of the entire EEG trace by an expert in pediatric EEG, blinded to the interpretation made at the bedside (gold standard).

Research hypothesis is that continuous neuromonitoring combining optimized quantitative EEG techniques and targeted advice from a neurophysiologist would allow the detection of a majority of seizure events requiring treatment and background trace abnormalities associated with critical encephalopathy.

ELIGIBILITY:
Inclusion Criteria :

* Patients younger than 2 years old hospitalized in the intensive care unit with an indication for neuromonitoring. The same patient may be included multiple times.
* Written non-opposition from legal representatives.
* Patients affiliated with or beneficiaries of a social security or similar scheme (CMU).

Exclusion Criteria :

* Parents who do not understand French.
* Inability to set up monitoring equipment (neurosurgery preventing access to electrode placement sites).
* Corrected age < 37 weeks of gestation (GA) for preterm infants.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients younger than 2 years old hospitalized in the intensive care unit with an indication for neuromonitoring
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance of neuromonitoring combining quantitative EEG and possible interpretation by a neurophysiologist in detecting neurological impairment. | 48 hours

SECONDARY OUTCOMES:
Evaluation of the detection of convulsive seizures | 48 hours
Evaluation of the classification of the background tracing in critical encephalopathy grade | 48 hours
Impact of tracing aids on intensivists' confidence level during decision-making | 48 hours
Number of suitable anticonvulsant treatments | 48 hours
Prescription period for anticonvulsant treatments | 48 hours
Hypothermia treatment rates indicated after subsequent rereading of the tracing by the expert | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided